CLINICAL TRIAL: NCT03892616
Title: Relative Bioavailability and Food Effect of a Single Dose of Different Solid Formulations of BI 1358894 Compared to a Single Dose of the Reference Tablet Formulation of BI 1358894 Following Oral Administration Under Fed and Fasted Conditions in Healthy Male Subjects (an Open-label, Single-dose, Randomised, Incomplete Blocks Crossover Design Study)
Brief Title: A Study in Healthy Men to Test if Taking Different Formulations of BI 1358894 With or Without Food Influences the Amount of BI 1358894 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1402-0010; 2018-003603-19 (EudraCT Number)
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — TRPC inhibitor BI 1358894; Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- TF1 fed (A)-TF2a fed (B)-TF2a fasted (C) (Experimental): 1 tablet of 100 milligram (mg) BI 1358894 was administrated as a single oral dose with 240 milliliter (mL) water 30 minutes (min) after a high-fat, high-calorie breakfast as treatment A (TF1; fed conditions) followed by a washout period of at least 17 days, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2a fed conditions) as treatment B followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 hours (h) (TF2a fasted conditions) as treatment C.
  Interventions: Drug: BI 1358894 (B); Drug: BI 1358894 (C); Drug: BI 1358894 (A)
- TF2b fed (D)-TF1 fed (A)-TF2a fed (B) (Experimental): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2b; fed conditions) as treatment D followed by at least 17 days of washout, followed by 1 tablet of 100 mg BI 1358894 was administrated as a single oral dose with 240mL water 30 min after a high-fat, high-calorie breakfast (TF1; fed conditions) as treatment A followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2a; fed conditions) as treatment B.
  Interventions: Drug: BI 1358894 (B); Drug: BI 1358894 (D); Drug: BI 1358894 (A)
- TF2b fasted (E)-TF2a fed (B)-TF1 fed (A) (Experimental): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2b; fasted conditions) as treatment E followed by washout period of at least 17 days, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2a; fed conditions) as treatment B followed by at least 17 days of washout, followed by 1 tablet of 100 mg BI 1358894 was administrated as a single oral dose with 240mL water 30 min after a high-fat, high-calorie breakfast (TF1; fed conditions) as treatment A.
  Interventions: Drug: BI 1358894 (B); Drug: BI 1358894 (E); Drug: BI 1358894 (A)
- TF2a fasted (C)- TF1 fed (A)-TF2b fed (D) (Experimental): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2a; fasted conditions) as treatment C followed by washout period of at least 17 days, followed by 1 tablet of 100 mg BI 1358894 was administrated as a single oral dose with 240mL water 30 min after a high-fat, high-calorie breakfast (TF1; fed conditions) as treatment A followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2b; fed conditions) as treatment D.
  Interventions: Drug: BI 1358894 (C); Drug: BI 1358894 (D); Drug: BI 1358894 (A)
- TF1 fed (A)- TF2b fasted (E)- TF2a fasted (C) (Experimental): 1 tablet of 100 mg BI 1358894 was administrated as a single oral dose with 240mL water 30 min after a high-fat, high-calorie breakfast (TF1; fed conditions) as treatment A followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2b; fasted conditions) as treatment E followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2a; fasted conditions) as treatment C.
  Interventions: Drug: BI 1358894 (C); Drug: BI 1358894 (E); Drug: BI 1358894 (A)
- TF2b fasted (E)-TF2b fed (D)- TF1 fed (A) (Experimental): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2b; fasted conditions) as treatment E followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2b; fed conditions) as treatment D followed by at least 17 days of washout, followed by 1 tablet of 100 mg BI 1358894 was administrated as a single oral dose with 240mL water 30 min after a high-fat, high-calorie breakfast (TF1; fed conditions) as treatment A.
  Interventions: Drug: BI 1358894 (D); Drug: BI 1358894 (E); Drug: BI 1358894 (A)
- TF2a fed (B)- TF2a fasted (C)-TF2b fed (D) (Experimental): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2a; fed conditions) as treatment B followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2a; fasted conditions) as treatment C followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2b; fed conditions) as treatment D.
  Interventions: Drug: BI 1358894 (B); Drug: BI 1358894 (C); Drug: BI 1358894 (D)
- TF2a fasted(C)-TF2b fasted(E)-TF2a fed(B) (Experimental): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2a; fasted conditions) as treatment C followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2b; fasted conditions) as treatment E followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2a; fed conditions) as treatment B.
  Interventions: Drug: BI 1358894 (B); Drug: BI 1358894 (C); Drug: BI 1358894 (E)
- TF2a fed(B)-TF2b fed(D)-TF2b fasted(E) (Experimental): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2a; fed conditions) as treatment B followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2b; fed conditions) as treatment D followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2b; fasted conditions) as treatment E.
  Interventions: Drug: BI 1358894 (B); Drug: BI 1358894 (D); Drug: BI 1358894 (E)
- TF2b fed(D)-TF2a fasted(C)-TF2b fasted(E) (Experimental): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2b; fed conditions) as treatment D followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2a; fasted conditions) as treatment C followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2b; fasted conditions) as treatment E.
  Interventions: Drug: BI 1358894 (C); Drug: BI 1358894 (D); Drug: BI 1358894 (E)
- TF2a fasted(C)-TF2a fed(B)-TF1 fed(A) (Experimental): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2a; fasted conditions) as treatment C followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2a; fed conditions) as treatment B followed by at least 17 days of washout, followed by 1 tablet of 100 mg BI 1358894 was administrated as a single oral dose with 240mL water 30 min after a high-fat, high-calorie breakfast (TF1; fed conditions) as treatment A.
  Interventions: Drug: BI 1358894 (B); Drug: BI 1358894 (C); Drug: BI 1358894 (A)
- TF1 fed (A)- TF2b fasted (E)-TF2b fed (D) (Experimental): 1 tablet of 100 mg BI 1358894 was administrated as a single oral dose with 240mL water 30 min after a high-fat, high-calorie breakfast (TF1; fed conditions) as treatment A followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2b; fasted conditions) as treatment E followed by at least 17 days of washout, followed by 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2b; fed conditions) as treatment D.
  Interventions: Drug: BI 1358894 (D); Drug: BI 1358894 (E); Drug: BI 1358894 (A)

INTERVENTIONS:
Drug: BI 1358894 (B) — Tablet formulation 2 (TF2a), fed
  Arms: TF1 fed (A)-TF2a fed (B)-TF2a fasted (C); TF2a fasted(C)-TF2a fed(B)-TF1 fed(A); TF2a fasted(C)-TF2b fasted(E)-TF2a fed(B); TF2a fed (B)- TF2a fasted (C)-TF2b fed (D); TF2a fed(B)-TF2b fed(D)-TF2b fasted(E); TF2b fasted (E)-TF2a fed (B)-TF1 fed (A); TF2b fed (D)-TF1 fed (A)-TF2a fed (B)
Drug: BI 1358894 (C) — Tablet formulation 2 (TF2a), fasted
  Arms: TF1 fed (A)- TF2b fasted (E)- TF2a fasted (C); TF1 fed (A)-TF2a fed (B)-TF2a fasted (C); TF2a fasted (C)- TF1 fed (A)-TF2b fed (D); TF2a fasted(C)-TF2a fed(B)-TF1 fed(A); TF2a fasted(C)-TF2b fasted(E)-TF2a fed(B); TF2a fed (B)- TF2a fasted (C)-TF2b fed (D); TF2b fed(D)-TF2a fasted(C)-TF2b fasted(E)
Drug: BI 1358894 (D) — Tablet formulation 2 (TF2b), fed
  Arms: TF1 fed (A)- TF2b fasted (E)-TF2b fed (D); TF2a fasted (C)- TF1 fed (A)-TF2b fed (D); TF2a fed (B)- TF2a fasted (C)-TF2b fed (D); TF2a fed(B)-TF2b fed(D)-TF2b fasted(E); TF2b fasted (E)-TF2b fed (D)- TF1 fed (A); TF2b fed (D)-TF1 fed (A)-TF2a fed (B); TF2b fed(D)-TF2a fasted(C)-TF2b fasted(E)
Drug: BI 1358894 (E) — Tablet formulation 2 (TF2b), fasted
  Arms: TF1 fed (A)- TF2b fasted (E)- TF2a fasted (C); TF1 fed (A)- TF2b fasted (E)-TF2b fed (D); TF2a fasted(C)-TF2b fasted(E)-TF2a fed(B); TF2a fed(B)-TF2b fed(D)-TF2b fasted(E); TF2b fasted (E)-TF2a fed (B)-TF1 fed (A); TF2b fasted (E)-TF2b fed (D)- TF1 fed (A); TF2b fed(D)-TF2a fasted(C)-TF2b fasted(E)
Drug: BI 1358894 (A) — Tablet formulation 1 (TF1), fed
  Arms: TF1 fed (A)- TF2b fasted (E)- TF2a fasted (C); TF1 fed (A)- TF2b fasted (E)-TF2b fed (D); TF1 fed (A)-TF2a fed (B)-TF2a fasted (C); TF2a fasted (C)- TF1 fed (A)-TF2b fed (D); TF2a fasted(C)-TF2a fed(B)-TF1 fed(A); TF2b fasted (E)-TF2a fed (B)-TF1 fed (A); TF2b fasted (E)-TF2b fed (D)- TF1 fed (A); TF2b fed (D)-TF1 fed (A)-TF2a fed (B)

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of a single dose of BI 1358894 administered as tablet formulation 2 (TF2a, TF2b) under fasted conditions compared with the tablet formulation 1 (TF1) of BI 1358894 under fed conditions following oral administration and to investigate the effect of food on the exposure with TF2 (TF2a, TF2b).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests.
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception of the female partner, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device (IUD) that started at least 2 months prior to first study drug administration, or barrier method (e.g. diaphragm with spermicide)
  * Sexually abstinent
  * A vasectomy performed at least 1 year prior to screening (with medical assessment of the surgical success)
  * Surgically sterilised female partner (including hysterectomy, bilateral tubal occlusion or bilateral oophorectomy)

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* C-Reactive Protein (CRP) > upper limit of normal (ULN), erythrocyte sedimentation rate (ESR) ≥15 millimeters/h, liver or kidney parameter above ULN, or any other laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Any lifetime history of suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
* Any suicidal ideation of type 2 to 5 on the Columbia Suicidal Severity Rating scale (C-SSRS) in the past 12 months (i.e. active suicidal thought, active suicidal thought with method, active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, single-dose, randomized, incomplete blocks crossover design study in healthy male was to test if taking different tablet formulations (TF1, TF2a, and TF2b) of BI 1358894 with or without food influences the amount of BI 1358894 in the blood.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Treatment Period 1
Arm/Group | TF1 Fed (A)-TF2a Fed (B)-TF2a Fasted (C) | TF2b Fed (D)-TF1 Fed (A)-TF2a Fed (B) | TF2b Fasted (E)-TF2a Fed (B)-TF1 Fed (A) | TF2a Fasted (C)- TF1 Fed (A)-TF2b Fed (D) | TF1 Fed (A)- TF2b Fasted (E)- TF2a Fasted (C) | TF2b Fasted (E)-TF2b Fed (D)- TF1 Fed (A) | TF2a Fed (B)- TF2a Fasted (C)-TF2b Fed (D) | TF2a Fasted(C)-TF2b Fasted(E)-TF2a Fed(B) | TF2a Fed(B)-TF2b Fed(D)-TF2b Fasted(E) | TF2b Fed(D)-TF2a Fasted(C)-TF2b Fasted(E) | TF2a Fasted(C)-TF2a Fed(B)-TF1 Fed(A) | TF1 Fed (A)- TF2b Fasted (E)-TF2b Fed (D)
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | TF1 Fed (A)-TF2a Fed (B)-TF2a Fasted (C) | TF2b Fed (D)-TF1 Fed (A)-TF2a Fed (B) | TF2b Fasted (E)-TF2a Fed (B)-TF1 Fed (A) | TF2a Fasted (C)- TF1 Fed (A)-TF2b Fed (D) | TF1 Fed (A)- TF2b Fasted (E)- TF2a Fasted (C) | TF2b Fasted (E)-TF2b Fed (D)- TF1 Fed (A) | TF2a Fed (B)- TF2a Fasted (C)-TF2b Fed (D) | TF2a Fasted(C)-TF2b Fasted(E)-TF2a Fed(B) | TF2a Fed(B)-TF2b Fed(D)-TF2b Fasted(E) | TF2b Fed(D)-TF2a Fasted(C)-TF2b Fasted(E) | TF2a Fasted(C)-TF2a Fed(B)-TF1 Fed(A) | TF1 Fed (A)- TF2b Fasted (E)-TF2b Fed (D)
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | TF1 Fed (A)-TF2a Fed (B)-TF2a Fasted (C) | TF2b Fed (D)-TF1 Fed (A)-TF2a Fed (B) | TF2b Fasted (E)-TF2a Fed (B)-TF1 Fed (A) | TF2a Fasted (C)- TF1 Fed (A)-TF2b Fed (D) | TF1 Fed (A)- TF2b Fasted (E)- TF2a Fasted (C) | TF2b Fasted (E)-TF2b Fed (D)- TF1 Fed (A) | TF2a Fed (B)- TF2a Fasted (C)-TF2b Fed (D) | TF2a Fasted(C)-TF2b Fasted(E)-TF2a Fed(B) | TF2a Fed(B)-TF2b Fed(D)-TF2b Fasted(E) | TF2b Fed(D)-TF2a Fasted(C)-TF2b Fasted(E) | TF2a Fasted(C)-TF2a Fed(B)-TF1 Fed(A) | TF1 Fed (A)- TF2b Fasted (E)-TF2b Fed (D)
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | TF1 Fed (A)-TF2a Fed (B)-TF2a Fasted (C) | TF2b Fed (D)-TF1 Fed (A)-TF2a Fed (B) | TF2b Fasted (E)-TF2a Fed (B)-TF1 Fed (A) | TF2a Fasted (C)- TF1 Fed (A)-TF2b Fed (D) | TF1 Fed (A)- TF2b Fasted (E)- TF2a Fasted (C) | TF2b Fasted (E)-TF2b Fed (D)- TF1 Fed (A) | TF2a Fed (B)- TF2a Fasted (C)-TF2b Fed (D) | TF2a Fasted(C)-TF2b Fasted(E)-TF2a Fed(B) | TF2a Fed(B)-TF2b Fed(D)-TF2b Fasted(E) | TF2b Fed(D)-TF2a Fasted(C)-TF2b Fasted(E) | TF2a Fasted(C)-TF2a Fed(B)-TF1 Fed(A) | TF1 Fed (A)- TF2b Fasted (E)-TF2b Fed (D)
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Met discontinuation criterion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | TF1 Fed (A)-TF2a Fed (B)-TF2a Fasted (C) | TF2b Fed (D)-TF1 Fed (A)-TF2a Fed (B) | TF2b Fasted (E)-TF2a Fed (B)-TF1 Fed (A) | TF2a Fasted (C)- TF1 Fed (A)-TF2b Fed (D) | TF1 Fed (A)- TF2b Fasted (E)- TF2a Fasted (C) | TF2b Fasted (E)-TF2b Fed (D)- TF1 Fed (A) | TF2a Fed (B)- TF2a Fasted (C)-TF2b Fed (D) | TF2a Fasted(C)-TF2b Fasted(E)-TF2a Fed(B) | TF2a Fed(B)-TF2b Fed(D)-TF2b Fasted(E) | TF2b Fed(D)-TF2a Fasted(C)-TF2b Fasted(E) | TF2a Fasted(C)-TF2a Fed(B)-TF1 Fed(A) | TF1 Fed (A)- TF2b Fasted (E)-TF2b Fed (D)
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all subjects who were randomized and treated with at least 1 dose of trial medication. The TS was used for the presentation of demographic and baseline characteristics and for the safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | TF1 Fed (A)-TF2a Fed (B)-TF2a Fasted (C) | TF2b Fed (D)-TF1 Fed (A)-TF2a Fed (B) | TF2b Fasted (E)-TF2a Fed (B)-TF1 Fed (A) | TF2a Fasted (C)- TF1 Fed (A)-TF2b Fed (D) | TF1 Fed (A)- TF2b Fasted (E)- TF2a Fasted (C) | TF2b Fasted (E)-TF2b Fed (D)- TF1 Fed (A) | TF2a Fed (B)- TF2a Fasted (C)-TF2b Fed (D) | TF2a Fasted(C)-TF2b Fasted(E)-TF2a Fed(B) | TF2a Fed(B)-TF2b Fed(D)-TF2b Fasted(E) | TF2b Fed(D)-TF2a Fasted(C)-TF2b Fasted(E) | TF2a Fasted(C)-TF2a Fed(B)-TF1 Fed(A) | TF1 Fed (A)- TF2b Fasted (E)-TF2b Fed (D) | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (12.0) | 46.0 (2.8) | 43.0 (7.1) | 46.0 (0.0) | 41.0 (11.3) | 46.5 (0.7) | 33.0 (18.4) | 46.0 (5.7) | 48.5 (2.1) | 35.5 (20.5) | 35.5 (10.6) | 47.0 (4.2) | 42.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Concentration of BI 1358894 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1358894 in plasma (Cmax).
Time Frame: Within 2 hours (h) before and at 10 minutes (min), 20min, 30min, 1h, 1h30min, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 48h, 72h, 96h, 144h, 192h, 240h, 312h after drug administration in each treatment period.
Population: Pharmacokinetic (PK) parameter analysis set (PKS) included all subjects in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: Nanomole (nmol) / Litre (L)
Groups:
- TF1 Fed (A): 1 tablet of 100 milligram (mg) BI 1358894 was administrated as a single oral dose with 240 milliliter (mL) water 30 min after a high-fat, high-calorie breakfast (Tablet formulation 1 (TF1); fed conditions) as treatment A.
- TF2a Fed (B): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2a; fed conditions) as treatment B.
- TF2a Fasted (C): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 hours (h) (TF2a; fasted conditions) as treatment C.
- TF2b Fed (D): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water 30 min after a high-fat, high-calorie breakfast (TF2b; fed conditions) as treatment D.
- TF2b Fasted (E): 2 tablets of 50mg BI 1358894 (total: 100mg) administrated as a single oral dose with 240 mL water after an overnight fast of at least 10 h (TF2b; fasted conditions) as treatment E.
Arm/Group | TF1 Fed (A) | TF2a Fed (B) | TF2a Fasted (C) | TF2b Fed (D) | TF2b Fasted (E)
Number analyzed (Participants) | 16 | 14 | 14 | 14 | 13
Nanomole (nmol) / Litre (L) | 497 (1.07) | 556 (1.08) | 484 (1.08) | 604 (1.08) | 909 (1.08)
Statistical Analysis 1: Comparison: TF1 Fed (A) vs TF2a Fasted (C); Relative bioavailability: ratio of adjusted geometric means was calculated using an analysis of variance (ANOVA). The model on logarithmic scale included random effect of 'subjects within sequences' and fixed effect of 'sequence or block', 'period', 'treatment'; Test type: Other; Ratio of adjusted geometric means [%] = 97.4, 90% CI 2-sided [82.3 to 115.3] — The ratio was calculated as adjusted geometric mean of TF2a fasted (C) as numerator and adjusted geometric mean of TF1 fed (A) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 25.44
Statistical Analysis 2: Comparison: TF1 Fed (A) vs TF2b Fasted (E); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 183.0, 90% CI 2-sided [154.0 to 217.4] — The ratio was calculated as adjusted geometric mean of TF2b fasted (E) as numerator and adjusted geometric mean of TF1 fed (A) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 25.44
Statistical Analysis 3: Comparison: TF2a Fed (B) vs TF2a Fasted (C); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 114.8, 90% CI 2-sided [96.5 to 136.6] — The ratio was calculated as adjusted geometric mean of TF2a fed (B) as numerator and adjusted geometric mean of TF2a fasted (C) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 25.44
Statistical Analysis 4: Comparison: TF2b Fed (D) vs TF2b Fasted (E); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 66.5, 90% CI 2-sided [55.5 to 79.5] — The ratio was calculated as adjusted geometric mean of TF2b fed (D) as numerator and adjusted geometric mean of TF2b fasted (E) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 25.44

2. Primary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) parameter analysis set (PKS) included all subjects in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Only participants with available PK data are included in the analysis.
Measure: Geometric Mean (Standard Error); unit: Nanomole (nmol)*hours(h)/Litre(L)
Arm/Group | TF1 Fed (A) | TF2a Fed (B) | TF2a Fasted (C) | TF2b Fed (D) | TF2b Fasted (E)
Number analyzed (Participants) | 16 | 14 | 14 | 13 | 13
Nanomole (nmol)*hours(h)/Litre(L) | 17695 (1.04) | 18934 (1.04) | 10645 (1.04) | 19356 (1.04) | 12655 (1.04)
Statistical Analysis 1: Comparison: TF1 Fed (A) vs TF2a Fasted (C); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 60.2, 90% CI 2-sided [55.3 to 65.5] — The ratio was calculated as adjusted geometric mean of TF2a fasted (C) as numerator and adjusted geometric mean of TF1 fed (A) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 12.65
Statistical Analysis 2: Comparison: TF1 Fed (A) vs TF2b Fasted (E); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 71.5, 90% CI 2-sided [65.6 to 78.0] — The ratio was calculated as adjusted geometric mean of TF2b fasted (E) as numerator and adjusted geometric mean of TF1 fed (A) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 12.65
Statistical Analysis 3: Comparison: TF2a Fed (B) vs TF2a Fasted (C); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 177.9, 90% CI 2-sided [162.8 to 194.3] — The ratio was calculated as adjusted geometric mean of TF2a fed (B) as numerator and adjusted geometric mean of TF2a fasted (C) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 12.65
Statistical Analysis 4: Comparison: TF2b Fed (D) vs TF2b Fasted (E); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 152.9, 90% CI 2-sided [139.5 to 167.7] — The ratio was calculated as adjusted geometric mean of TF2b fed (D) as numerator and adjusted geometric mean of TF2b fasted (E) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 12.65

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Error); unit: Nanomole (nmol)*hours(h)/Litre(L)
Arm/Group | TF1 Fed (A) | TF2a Fed (B) | TF2a Fasted (C) | TF2b Fed (D) | TF2b Fasted (E)
Number analyzed (Participants) | 16 | 14 | 14 | 13 | 13
Nanomole (nmol)*hours(h)/Litre(L) | 19425 (1.04) | 20596 (1.04) | 11715 (1.04) | 20752 (1.05) | 13818 (1.05)
Statistical Analysis 1: Comparison: TF1 Fed (A) vs TF2a Fasted (C); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 60.3, 90% CI 2-sided [55.4 to 65.7] — The ratio was calculated as adjusted geometric mean of TF2a fasted (C) as numerator and adjusted geometric mean of TF1 fed (A) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 12.70
Statistical Analysis 2: Comparison: TF1 Fed (A) vs TF2b Fasted (E); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 71.1, 90% CI 2-sided [65.2 to 77.6] — The ratio was calculated as adjusted geometric mean of TF2b fasted (E) as numerator and adjusted geometric mean of TF1 fed (A) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 12.70
Statistical Analysis 3: Comparison: TF2a Fed (B) vs TF2a Fasted (C); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 175.8, 90% CI 2-sided [160.8 to 192.2] — The ratio was calculated as adjusted geometric mean of TF2a fed (B) as numerator and adjusted geometric mean of TF2a fasted (C) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 12.70
Statistical Analysis 4: Comparison: TF2b Fed (D) vs TF2b Fasted (E); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 150.2, 90% CI 2-sided [136.9 to 164.7] — The ratio was calculated as adjusted geometric mean of TF2b fed (D) as numerator and adjusted geometric mean of TF2b fasted (E) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 12.70

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over the Time Interval From 0 to 72 Hours (AUC0-72)
Description: Area under the concentration-time curve of BI 1358894 in plasma over the time interval from 0 to 72 hours (AUC0-72).
Time Frame: Within 2 hours (h) before and at 10 minutes (min), 20min, 30min, 1h, 1h30min, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 48h, 72h after drug administration in each treatment period.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: Nanomole (nmol) * hours (h) / Litre (L)
Arm/Group | TF1 Fed (A) | TF2a Fed (B) | TF2a Fasted (C) | TF2b Fed (D) | TF2b Fasted (E)
Number analyzed (Participants) | 16 | 14 | 14 | 14 | 13
Nanomole (nmol) * hours (h) / Litre (L) | 11742 (1.04) | 12297 (1.05) | 6635 (1.05) | 13109 (1.05) | 8273 (1.05)
Statistical Analysis 1: Comparison: TF1 Fed (A) vs TF2a Fasted (C); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 56.5, 90% CI 2-sided [51.8 to 61.7] — The ratio was calculated as adjusted geometric mean of TF2a fasted (C) as numerator and adjusted geometric mean of TF1 fed (A) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 13.02
Statistical Analysis 2: Comparison: TF1 Fed (A) vs TF2b Fasted (E); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 70.5, 90% CI 2-sided [64.4 to 77.1] — The ratio was calculated as adjusted geometric mean of TF2b fasted (E) as numerator and adjusted geometric mean of TF1 fed (A) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 13.02
Statistical Analysis 3: Comparison: TF2a Fed (B) vs TF2a Fasted (C); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 185.3, 90% CI 2-sided [169.4 to 202.8] — The ratio was calculated as adjusted geometric mean of TF2a fed (B) as numerator and adjusted geometric mean of TF2a fasted (C) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 13.02
Statistical Analysis 4: Comparison: TF2b Fed (D) vs TF2b Fasted (E); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 158.4, 90% CI 2-sided [144.3 to 173.9] — The ratio was calculated as adjusted geometric mean of TF2b fed (D) as numerator and adjusted geometric mean of TF2b fasted (E) as denominator, *100. Intra-individual geometric coefficient of variation (gCV [%]) = 13.02

ADVERSE EVENTS:
Time Frame: From drug administration until the next drug administration, or until the end of the trial, up to 22 days.
Description: The treated set (TS) included all subjects who were randomized and treated with at least 1 dose of trial medication. The TS was used for the presentation of demographic and baseline characteristics and for the safety analyses.
Arm/Group | TF1 Fed (A) | TF2a Fed (B) | TF2a Fasted (C) | TF2b Fed (D) | TF2b Fasted (E)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14 | 0/14 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/14 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 7/16 | 9/14 | 10/14 | 7/14 | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TF1 Fed (A) (N=16) | TF2a Fed (B) (N=14) | TF2a Fasted (C) (N=14) | TF2b Fed (D) (N=14) | TF2b Fasted (E) (N=13)
Headache (Nervous system disorders) | 5 | 6 | 5 | 6 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT03892616/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT03892616/SAP_001.pdf